CLINICAL TRIAL: NCT02775370
Title: Phase II Study of Apatinib Mesylate Administered as a Daily Oral Treatment in Patients With Recurrent/Metastatic Adenoid Cystic Carcinoma of the Head and Neck
Brief Title: A Study of Apatinib in Recurrent/Metastatic Adenoid Cystic Carcinoma of the Head and Neck
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, M.D., Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016HNRT003
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib group (Experimental): Apatinib Mesylate administered as a daily oral treatment
  Interventions: Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Apatinib Mesylate — Apatinib Mesylate will be administered orally at 500 mg once daily for 5 consecutive days, and this was followed by a 2-day rest every week; each cycle consisted of 28 days

SUMMARY:
This is a non-randomized, phase II, open label study of Apatinib Mesylate in patients with Head and neck recurrent/metastatic adenoid cystic carcinoma (ACC). The primary purpose of this study is to evaluate the efficacy and safety of Apatinib Mesylate in patients with ACC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenoid cystic carcinoma
2. Recurrent/Metastatic disease documented as having shown progression on a scan (CT, MRI) compared to a previous scan taken at any time in the past. Progression must be documented according to RECIST criteria.
3. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria
4. Disease that is not amenable to surgery, radiation or combined modality therapy with curative intent and was previously treated with chemotherapy
5. 18 years or older
6. Karnofsky score over 60
7. Previous treatment with chemotherapy, targeted agents, loco-regional therapy (e.g. chemoembolization) are permitted providing that toxicity has resolved to < or = grade 1 at study entry and that last treatment was at least 4 weeks prior to baseline assessment.
8. Adequate organ function
9. A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
10. A patient who signed the informed consent prior to the participation of the study and who understands that he or she has a right to withdrawal from participation in the study at any time without any disadvantages.

Exclusion Criteria:

1. A patient with no measurable disease
2. Prior chemotherapy, radiation therapy or surgery within 4 weeks prior to study entry except palliative radiotherapy to non-target lesions (within 2 weeks prior to study entry)
3. A patient with previous active or passive immunotherapy
4. A patient with intestinal obstruction or impending obstruction, recent active upper GI bleeding
5. A pregnant or lactating patient
6. A patient of childbearing potential without being tested for pregnancy at baseline or with being tested for positive. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential)
7. A man or woman of childbearing potential who has no willingness to use a contraceptive measure during the study
8. A patient with history of another malignant disease within past 5 years, except curatively treated basal cell carcinoma of skin and cervical carcinoma in situ.
9. A patient with history of uncontrolled seizures, central nervous system disorder or psychiatric disorders that are considered clinically significant by the investigator that would prohibit the understanding of informed consent or that may be considered to interfere with the compliance of the administration of the study medications.
10. A patient with clinically significant heart disease (e.g. congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmia, etc) or myocardial infarction within past 12 months.
11. Ongoing cardiac arrhythmia of grade > or = 2, atrial fibrillation of any grade, or QTc interval > 450 msec for males or > 470 msec for female.
12. A patient with interstitial pneumonia or diffuse symptomatic fibrosis of the lungs
13. A patient with organ transplantation requiring immunosuppressive therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 6 months
  To determine 6 month PFS of Apatinib Mesylate when administered as monotherapy in patients with metastatic adenoid cystic carcinoma

SECONDARY OUTCOMES:
Overall survival rate | 2 years
  from date of enrollment until date of first death from any cause, assessed up to 2 years
Response rate | 8 weeks
  CT scan will be evaluated every 2 cycles (per 8 weeks)till progression. Response rate will be evaluated by RECIST criteria
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chenping Zhang, M.D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University; Guopei Zhu, M.D., Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai ninth people's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ye L, Zhang L, Li R, Pan X, Li J, Dou S, Jiang W, Wang C, Chen W, Zhu G. Combined all-trans retinoic acid with low-dose apatinib in treatment of recurrent/metastatic head and neck adenoid cystic carcinoma: A single-center, secondary analysis of a phase II study. Cancer Med. 2023 Apr;12(8):9144-9155. doi: 10.1002/cam4.5653. Epub 2023 Feb 3. PMID 36734294
- [Derived] Zhu G, Zhang L, Dou S, Li R, Li J, Ye L, Jiang W, Dong M, Ruan M, Yang W, Zhang C. Apatinib in patients with recurrent or metastatic adenoid cystic carcinoma of the head and neck: a single-arm, phase II prospective study. Ther Adv Med Oncol. 2021 May 8;13:17588359211013626. doi: 10.1177/17588359211013626. eCollection 2021. PMID 33995600